CLINICAL TRIAL: NCT06401655
Title: A Pilot Study About Financial Coaching for Adults Living With Acquired Brain Injury
Brief Title: Financial Coaching for Adults Living With Acquired Brain Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Lisa Engel, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS26252 (H2023:356)
Record Dates: First submitted 2024-04-30; First posted 2024-05-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Brain Injuries; Stroke
Keywords: Financial capability; Financial management; Financial self-efficacy; Goal attainment; Strategy Training
MeSH Terms: conditions — Brain Injuries; Stroke

STUDY DESIGN:
Intervention Model Description: This pilot study will utilize a longitudinal concurrent mixed-methods research design that gathers and analyzes qualitative and quantitative data overtime about a new 10-session financial coaching program the investigators have developed. The data collected will be used to inform improvements to future related studies and programs for people living with brain injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (pilot) (Experimental): The total time in this study for an ABI-survivor participant is 10 hours and 15 minutes which includes 7.5 hours of intervention time and 2.75 hours of data collection time.
  This is an individualized, in-person 10-session financial coaching intervention program. Each session is 45-minutes. In total, participants will be asked to participate in up to 7 hours and 30 minutes of intervention time with a trained Occupational Therapist. Each session will happen 1-1.5 weeks apart and the financial coaching program will last over 3-4 months. The financial coaching sessions will only be offered in-person (at MBIA Winnipeg location, in their home, at the University of Manitoba/Banntyne Campus, or other community locations acceptable/consented by the participant).
  Interventions: Behavioral: Financial Coaching for People living with Acquired Brain Injury (FC-ABI)

INTERVENTIONS:
Behavioral: Financial Coaching for People living with Acquired Brain Injury (FC-ABI) — This is an individualized, in-person 10-session financial coaching intervention program. Each session is 45-minutes. In total, participants will be asked to participate in up to 7 hours and 30 minutes of intervention time with a trained Occupational Therapist. Each session will happen 1-1.5 weeks apart and the financial coaching program will last over 3-4 months. The financial coaching sessions will only be offered in-person (at MBIA Winnipeg location, in their home, at the University of Manitoba/Banntyne Campus, or other community locations acceptable/consented by the participant).

SUMMARY:
This pilot study will utilize a longitudinal concurrent mixed-methods research design that gathers and analyzes qualitative and quantitative data overtime about a new 10-session financial coaching program the investigators have developed. The data collected will be used to inform improvements to future related studies and programs for people living with acquired brain injury (ABI).

These mixed-methods data from each method will be integrated to provide a comprehensive understanding of the intervention (i.e., the financial coaching program). Each individualized intervention per ABI-survivor participant will be completed over 3-4 months (i.e., 12-14 weeks).

DETAILED DESCRIPTION:
The people to be recruited in the study include:

1. Adults living with acquired brain injuries (ABI; "ABI-survivor participant"), and
2. Close or trusted others of the adult participants who live with ABI (involvement with the consent of the adult living with ABI; "Close-other support person").

The investigators will recruit participants through community partner organizations. The principal investigator (Dr. Engel) has established relationship with community organizations.

The primary participants for this study are adults who live with Acquired Brain Injury (ABI; i.e., ABI-survivor participants). However, with the consent and guidance of the ABI-survivor participants, the investigators will invite up to one close-other (e.g., caregiver, family, involved friend) of the ABI-survivor participant to take part in the study as a support-person in the intervention with the ABI-survivor participant (involvement of close-others is described more below).

The investigators will recruit up to five ABI-survivors (n=5), each who may or may not have a support person involved in the study. This sample size will be sufficient to generate required information for the study aim and objectives, as there will be some homogeneity to the sample (i.e., adults living with ABI) while also looking for heterogeneity in other participant qualities (i.e., gender, age, time since first brain injury).

The total time in this study for an ABI-survivor participant is 10 hours and 15 minutes which includes 7.5 hours of intervention time and 2.75 hours of data collection time.

This is an individualized, in-person 10-session financial coaching intervention program. Each session is 45-minutes. In total, participants will be asked to participate in up to 7 hours and 30 minutes of intervention time with a trained Occupational Therapist. Each session will happen 1-1.5 weeks apart and the financial coaching program will last over 3-4 months.

The Financial Coaching Program (FCp) will consist of 10 sessions that will last 45-minutes per session. Each session will be in a 1:1 format with the participant and financial coach (i.e., interventionist) who is a trained and registered Occupational Therapist. Participants are welcome to invite a close other (e.g., family, caregiver, friend) to attend and participate in sessions as a support person and as agreed upon during informed consent and while getting started in the study; although, at any time the participant can choose to not include or stop including their close other for some or all of the remaining FCp sessions.

FCp sessions will take place in a variety of spaces, dependent on the participant's preference. Sessions can be completed in the participant's home, the meeting spaces of the Manitoba Brain Injury Association, or office space in the College of Rehabilitation Science building. Sessions can take place in another community space if requested by the participant.

The FCp will follow a Cognitive Orientation to daily Occupational Performance (CO-OP) format. The CO-OP method will focus on building skills through the development and use of cognitive strategies. These problem-solving strategies can then be used to improve performance in other aspects of daily life and in new situations. The FCp financial coaches have been trained in CO-OP basics online course and completed the certificate consolidation course.

During the FCp sessions, the participant will work with a financial coach to practice problem solving skills and work toward achieving 3 financial goals: 2 of these goals will be addressed directly during multiple FCp sessions and 1 goal will be "unaddressed" or "untrained", only to be discussed in the last session related to generalization of learning to other goals. The financial coach will not instruct participants but will instead work collaboratively with them to develop strategies and action plans. The participant and financial coach will agree on homework assignments to complete between sessions, which will be reviewed at the beginning of each subsequent session.

The FCp will be facilitated by a financial coach (I.e, intervnetionists), who will be a paid research staff member and part of the research team identified in the informed consent forms. The financial coach is an occupational therapist with experience working with individuals with brain injury. The financial coaches hired for this study have completed the following additional training:

* Cognitive Orientation to Occupational Performance (CO-OP) comprehensive online course and completed the certificate consolidation
* SEED Financial Empowerment Program certificate training for financial literacy/capability facilitators (train-the-trainer program; https://seedwinnipeg.ca)
* Training through Prosper Canada Financial Empowerment Foundations

ELIGIBILITY:
Acquired Brain Injury (ABI-Survivor) Participants

The inclusion criteria for ABI-survivor participants are:

1. Age 18 years or older
2. Self-report living with ABI (e.g., traumatic brain injury, stroke, non-traumatic brain injury, or brain injury due to other mechanisms) and chronic/ongoing ABI related symptoms or changes.
3. Self-report to be at least 6 months since the last or only ABI incident (to ensure not in acute stage of brain injury recovery).
4. Currently living in Winnipeg, Manitoba (i.e., the city where the in-person intervention sessions will take place).
5. Can participate sessions that are up to 1-hour in length.
6. Can identify 3 financial-related goals they want to address during the study/financial coaching program over the next 3-4 months.
7. Are interested in wanting to address their financial-related goals with a trained Occupational Therapist.
8. Able to attend in-person sessions at various Winnipeg locations that are convenient for them and if transportation cost support is provided (e.g., parking costs, bus tickets, taxi costs).

The exclusion criteria for ABI-survivor participants are:

1. Are not able to participate in in-person sessions that are at least 45 minutes long.
2. Are not able to communicate in English (verbal & written)
3. Unable to complete informed consent and capacity check questions for this study (see informed consent forms).

As the investigators are only looking to recruit up to five (n=5) ABI-survivor participants for this study, during screening the investigators will use maximum variation sampling (a specific form of purposive sampling) to guide inclusion if more than five ABI-survivors express interest in this study and are eligible to participate. During screening, the investigators will ask people about self-identified gender in an open-ended question that the investigators then categorize (i.e., man, woman, non-binary) and age (i.e., 18-30 years old, 31-60 years old, greater than 60 years old). Age and gender have been noted to have an influence on financial capability and financial well-being.

Close-Other Support Persons

The inclusion criteria for the Close-Other Support Person are:

1. Be identified by the ABI-survivor participant as someone they would like to have involved in this intervention.
2. Be 18 years or older.
3. Live in Winnipeg, Manitoba or immediate surrounding environment.
4. Be willing and able to participate in at least 3 sessions in-person financial coaching intervention sessions with the ABI-survivor participant (with times and locations to be scheduled convenient to support-person, the ABI-survivor participant, and OT interventionist)

The exclusion criteria for the Close-Other Support Person are:

1. Are not able to participate in in-person sessions that are at least 45 minutes long.
2. Are not able to communicate in English (verbal & written)
3. Unable to complete informed consent and capacity check questions for this study (see informed consent forms).
4. The ABI-participant does not provide consent for this person to be a part of their intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | through study completion, an average 3 months
  COPM is a client-centred tool for individuals to identify and rank problems that restrict their participant in their daily life. Scale score 0-10 on satisfaction and 0-10 on performance of two study goals. Higher scores means more satisfaction or more self-perceived performance related to the goal.
Goal Attainment Scaling (GAS) | through study completion, an average 3 months
  Goal attainment scaling is a client-centred approach that makes it easier for clients to create personalized and relevant goals for therapy and tracks how far the intervention is moving in the direction of attaining the set goals. Scale of 1-5 for each goals, where 3 is equal to goal being met, 1-2 is goal progress but goal not met, and 4-5 is goal is met and exceeded.

SECONDARY OUTCOMES:
Financial Self Efficacy Scale (FSES) #1 - Rothwell | through study completion, an average 3 months
  FSES is a measure of an individual's skills, knowledge and ability to manage their household finance. Scale responses 4-20, with higher numbers indicating more financial self-efficacy.
Financial Self Efficacy Scale (FSES) #2 - Lown | through study completion, an average 3 months
  FSES was developed as a tool for researchers to measure how behavior financial management and a basis for understanding, motivating, and guiding clients. Scale 4-24, with higher scores indicating more financial self-efficacy.
InCharge Financial Distress/Well-being Scale- Prawitz | through study completion, an average 3 months
  The InCharge financial distress/financial well-being scale measure a latent construct representing one's financial state on a continuum ranging from distress or lowest level of financial well-being to no distress/highest level of financial well-being. Scale 8-80, with higher scores indicating less financial distress/more financial wellbeing.

OTHER OUTCOMES:
Qualitative interviews | through study completion, an average 3 months
  Explore the perspectives of people involved, including participants living with brain injury and close others/caregivers, and research staff who provided the program service (interventionists), about the financial coaching programs meaningfulness, usefulness, how to continue to improve the program.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Engel, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
No plan for sharing individual participant data to other researchers as dataset includes full qualitative interview transcripts which could identify participants if shared in entirety.